CLINICAL TRIAL: NCT03648216
Title: The Effect of Experimentally Increasing Sedentary Behaviour on Subjective Well-being in Non-sedentary University Students
Brief Title: The Effect of Experimentally Increasing Sedentary Behaviour on Subjective Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 112536
Record Dates: First submitted 2018-08-14; First posted 2018-08-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Lifestyle; Quality of Life
Keywords: Sedentary Behaviour; Subjective Well-Being; University Students
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Upon obtaining consent, eligible participants will complete a week-long baseline period and then will be randomly assigned to either a 1-week intervention or control group, followed by a 1-week follow-up period.
Who Masked: Participant
Masking Description: Study advertisements and information provided to participants will focus on non-specific behaviour change, in order to mask participants to the purpose of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a pedometer and HAPA behavioural counseling with the aim of limiting their daily step count to <5000 steps per day, over a one week period. Counseling strategies will be grounded in the HAPA model - specifically, creating an action plan and coping strategies for maximizing their daily sedentary behaviour and minimizing steps taken. Strategies may include: driving to locations more often, refraining from physical activity as much as possible, and/or completing tasks in sedentary postures.
  Interventions: Behavioral: HAPA behavioural counseling
- Control Group (No Intervention): The control group will not receive any behavioural intervention or instruction.

INTERVENTIONS:
Behavioral: HAPA behavioural counseling — Behavioural counseling grounded in the Health Action Process Approach (HAPA; i.e., action planning and coping planning) to maximize sedentary behaviour and minimize steps taken.
  Arms: Intervention Group

SUMMARY:
This study will explore the causality between outcomes of subjective well-being and sedentary behavior, through experimentally increasing the sedentary behavior levels of active university students. Half of the eligible participants will receive a behavioral counseling intervention to increase sedentary behavior over one week, while the other half will receive no instructions. After one week, all participants will receive no instructions and continue to wear the inclinometer for another week.

DETAILED DESCRIPTION:
The relationship between subjective well-being (SWB) and sedentary behavior (SB) has been briefly explored. However, the causality of the relationship (i.e., do higher levels of SB cause changes in SWB, or vice-versa) has not been fully examined. Experimentally increasing SB and observing the potential subsequent effect on SWB, in otherwise non-sedentary individuals, may help to determine the causation between SB and SWB.

An active sample of full-time university students attending Western University will be recruited. Upon obtaining consent, demographics will be taken. Baseline sedentary behavior levels will be confirmed objectively through inclinometer wear for 1-week. Upon confirmation of sufficient sedentary/non-sedentary time, participants will complete questionnaires assessing past-week: SWB, SB, physical activity, depression, and anxiety questionnaires. Participants will also be randomized to either a behavioral counseling intervention group, or a no-contact control group. Participants will then continue wearing the inclinometer for 1 week. After the intervention week, participants will complete the questionnaires again, after which all participants will be told to continue daily behavior, and wear the inclinometer for another week. Upon completion of this follow-up week, participants will complete questionnaires again.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Full-time student attending Western University
* Able to read and write in English
* Self-reporting ≥150 minutes/week of moderate-vigorous physical activity

Exclusion Criteria:

* Self-reporting a mental illness
* Currently having a physical disability that would prevent walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Change from pre-randomization Subjective Well-Being (Affect) at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Subjective Well-Being (specifically, affect) will be assessed through the Positive Affect & Negative Affect Scale (PANAS).
  The PANAS consists of a number of words that describe different feelings and emotions. Participants indicate the extent to which they feel a particular feeling and emotion over the past week, using a 5-point scale that ranges from 1 "very slightly or not at all" to 5 "extremely".
  An overall score for both positive and negative affect is calculated by summing up the points for those particular feelings/emotions (e.g., interested for positive affect, distressed for negative affect). Scores for positive affect can range from 10-50, with higher scores representing higher levels of positive affect. Scores for negative affect can range from 10-50, with lower scores representing lower levels of negative affect.
Change from pre-randomization Subjective Well-Being (Life Satisfaction) at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Subjective Well-Being (specifically, life satisfaction) will be assessed through the Satisfaction with Life Scale (SWLS); a 5-item scale designed to measure global cognitive judgments of one's life satisfaction.
  Participants indicate how much they agree or disagree with each of the 5-items over the past week, using a 7-point scale that ranges from 7 "strongly agree" to 1 "strongly disagree". An overall score (from 5 to 35) is calculated through summing the responses to the 5-items.
  Recommended cutoffs for interpretation are: 5-9, extremely dissatisfied; 10-14, dissatisfied; 15-19, slightly dissatisfied; 20, neutral; 21-25, slightly satisfied; 26-30, satisfied; 31-35, very satisfied.
Change from pre-randomization Subjective Well-Being (Eudaimonic Well-Being) at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Subjective Well-Being (Eudaimonic Well-Being) will be assessed through the Subjective Vitality Scale (SVS); a 6- or 7-item scale that assesses the state of feeling alive and alert - to having energy available to the self. For the purposes of this study, the 6-item individual difference level version of the SVS will be utilized.
  Participants indicate the degree in which a statement/item is true in general in their life, ranging from 1 "not at all" to 7 "very true". An overall score is obtained by averaging the scores for each of the 6-items, with higher scores indicating a greater feeling of vitality.
Change from pre-randomization Subjective Well-Being at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Subjective Well-Being will be assessed through the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).
  The WEMWBS consists of 14-items that assesses subjective well-being through both hedonic and eudaimonic dimensions of well-being. Participants select the option that best describes their experience with each of the 14-items over the last week (note: the original questionnaire assesses the last two weeks), using a 5-point scale that ranges from 1 "none of the time" to 5 "all of the time".
  A total score is calculated by summing the 14 individual statement scores. The minimum score is 14 and the maximum is 70, with higher scores indicating greater levels of subjective well-being.

SECONDARY OUTCOMES:
Change from pre-randomization self-reported Physical Activity at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Average self-reported total weekday and weekend time spent in moderate and vigorous physical activities in the last 7 days will be assessed through the International Physical Activity Questionnaire Seven - Short Form Past 7 Days (IPAQ-S7S).
  Participants report how many days per week (0-7) and how many hours/minutes per day they spent engaged in vigorous and moderate intensity physical activity, as well as walking.
Change from pre-randomization self-reported Sedentary Behaviour at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Average self-reported weekday and weekend domain-specific time spent sedentary over the past 7 days will be assessed through the modified SIT-Q 7d questionnaire. Participants indicate on a scale of responses the range of times that best correspond to the average amount of time they spent sedentary on weekdays/weekends in domains of: Sleeping and Napping, Meals, Transportation, Occupation(s), Screen Time, and Other Activities, during the past 7 days. Response ranges typically span 30 minutes to 1 hour (e.g., Less than 30 minutes, 1-2 hours).
  Average total sitting time per weekday will be assessed through a single question on the International Physical Activity Questionnaire Seven - Short Form Past 7 Days (IPAQ-S7S): "During the last 7 days, how much time did you spend sitting on a weekday?" Average total sitting time per day; assessed through the International Physical Activity Questionnaire Seven - Short Form Past 7 Days (IPAQ-S7S)
Change from pre-randomization Depression at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Depressive symptomatology will be assessed through the Centre for Epidemiological Studies Depression Scale (CES-D).
  The CES-D scale is a short self-report scale designed to measure depressive symptomatology in the general population. Participants indicate how often in the past week they have felt or behaved for each of the 20 feelings/behaviors in the scale. Options range from: rarely or none of the time (less than 1 day), some or little of the time (1-2 days), occasionally or a moderate amount of time (3-5 days), and most or all of the time (5-7 days). These options correspond to a score of either: 0, 1, 2, or 3, depending on the framing of the question.
  A total score is achieved through summing the scores for all 20 questions; scores range from 0-60, with lower scores indicating a lower symptomatomology for depression. A clinical cut-off point of 20 has been recommended.
Change from pre-randomization Anxiety (State) at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  State anxiety will be assessed through the State-Trait Anxiety Inventory (STAI) Form Y-1. Participants read each of the 20 statements and then write the number in the blank at the end of the statement that indicates how they feel right now (i.e., at this moment).
  Responses range from: 1 - not at all, to 4 - very much so; these response correspond to a score of 1-4 for anxiety-related items, and 4-1 for anxiety-absent items. A total score is obtained by summing the scores for each question. Total scores range from 20-80, with higher scores indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the State Anxiety scale.
Change from pre-randomization objectively-measured Sedentary Behaviour at 1-week post-intervention and 1-week follow-up | Baseline, 1-week post-intervention, and 1-week follow-up
  Average objectively-reported weekday and weekend time spent sedentary over the past 7 days will be assessed through the ActivPAL4 inclinometer. Participants will wear the device on their thigh for a period of 7 days. The inclinometer is able to track and distinguish between sitting, standing, and other non-sedentary behaviours. The ActivPAL software can be used to extract data from the device to form daily levels of sedentary behaviour over the last 7 days. Activity can then be averaged to form a weekly average of time spent sedentary.

OTHER OUTCOMES:
Age | Baseline
  Assessed with a single-item question: "What is your age?"
Gender | Baseline
  Assessed with a single-item question: "What is your preferred gender?"
Program of Study | Baseline
  Assessed with a single-item question: "What is your current program of study?"
Year of Study | Baseline
  Assessed with a single-item question: "What is your current year of study?"
Degree Pursuing | Baseline
  Assessed with a single-item question: "What degree are you pursuing?"
Ethnicity | Baseline
  Assessed with a single-item question: "Which ethnicity do you most closely identify with?"

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — Western University
Locations (1):
- Exercise and Health Psychology Lab, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the research results, IPD will be shared into the Federated Research Data Repository (FRDR)
Supporting Information: Study Protocol
Time Frame: Data will become available upon publication of the research results, and will be available for 5 years after depositing.
Access Criteria: Members of the FRDR will be able to access the data.
URL: http://www.frdr.ca/repo/?locale=en